CLINICAL TRIAL: NCT06586190
Title: Outpatient Floor Pedal Bike Utilization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00101617
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-06

CONDITIONS: Femur Fracture; Tibia Fracture; Ankle Injuries
Keywords: floor pedal bike; lower extremity; rehabilitation
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures; Ankle Injuries | interventions — Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Arm (Other): Patients with lower extremity traumatic injuries that are medically clear for physically ready for therapy and will receive a floor pedal bike with guided exercises at home.
  Interventions: Other: Floor Pedal Bike with Guided Instructions for Home

INTERVENTIONS:
Other: Floor Pedal Bike with Guided Instructions for Home — Patients with lower extremity traumatic injuries that are medically clear for physically ready for therapy and will receive a floor pedal bike with guided exercises at home.

SUMMARY:
The goals of this clinical trial are: to test the feasibility of identifying patients and getting patients the floor pedal bikes, to test how well floor pedal bikes help patients with lower body injuries heal, and to test methods of patient self-reported logs for home pedal bike use.

Participants will be given a floor pedal bike at first post-operative appointment where weightbearing restrictions are lifted (weight-bearing as tolerated) along with instructions on utilization. Participants will be asked to complete patient reported outcome measure surveys at each follow-up visit.

DETAILED DESCRIPTION:
The goals of this clinical trial are:

1. to test the feasibility of identifying patients and getting patients the floor pedal bikes themselves
2. to test the efficacy of floor pedal bikes in the rehabilitation of patients with lower extremity orthopedic trauma injuries without formal physical therapy or as a supplement to preexisting and/or future physical therapy. We hope that these bikes will either supplement patient's preexisting therapy or allow them to complete therapy at home if they are unable to obtain formal physical therapy and
3. to test various methods of patient self-reported logs for home pedal bike utilization, whether electronic or hard paper copy.

Participants will be given a floor pedal bike at first post-operative appointment where weightbearing restrictions are lifted (weight-bearing as tolerated) along with instructions on utilization. Participants will be asked to complete patient reported outcome measure surveys at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Operative fractures of the femur, tibia and select ankle injuries
* Under the care of an orthopaedic surgeon
* English or Spanish competent
* 12 month follow up

Exclusion Criteria:

* Type IIIB/C fracture
* Unable to provide consent/need for an LAR
* Major lower extremity peripheral nerve injury (ex. foot drop, sciatic nerve palsy, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Return to Work/Functional Activity | Baseline, 3, 6, 12 months
  The primary assessment tool will be the International Physical Activity Questionnaire.
  IPAQ measures the total amount of physical activity completed in a 7 day period by calculating the minutes per week in in each physical activity level domain (walking, moderate and vigorous) by a metabolic equivalent energy (MET) expenditure estimate.
  Walking = 3.3 x number of walking minutes x number of walking days Moderate activity= 4.0 x number activity minutes x number of days Vigorous activity = 8 x number of activity minutes x number of days Total = Walking MET-min/wk+moderate MET-min/wk+vigorous MET-min/wk

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | Baseline, 3, 6, 12 months
  Scores range between 0-100. Higher scores indicate higher resilience.
Tampa Scale for Kinesiophobia (TSK) | Baseline, 3, 6, 12 months
  This scale is 17 items and uses a 4-point Likert scale ranging from 'strongly disagree' to 'strongly agree'. The TSK is a validated measure for surgical and musculoskeletal patients. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Pain Catastrophizing Scale (PCS) | Baseline, 3, 6, 12 months
  Scores range between 0-52. A higher score indicates a greater degree or pain catastrophizing.
Veterans RAND 12 Item Health Survey (VR-12) | Baseline, 3, 6, 12 months
  Patients will complete the Veterans RAND 12 Item Health Survey (VR12).The VR-12 is a measure of global health that corresponds to seven domains: general health, physical functioning, role limitations, pain, fatigue, social functioning, and mental health. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
PROMIS Pain Interference Short Form | 3, 6, 12 months
  Scores range from 8 to 40. A higher score indicates greater pain interference.
PROMIS Physical Function Short Form | 3, 6, 12 months
  T-scores range from 14.1 to 61.7. T-scores of 14.1-30.0 represent severe impairment, 30.0-40.0 represent moderate impairment, 40.0-45.0 represent mild impairment, and 45.0-61.7 indicate no impairment
Brief Pain Inventory (BPI) | 3, 6, 12 months
  The BPI is a commonly used and validated 15-item measure of pain intensity and interference with daily life. Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Performance test - Timed up and go test | 3, 6, 12 months
  Participants begin in a seated position. They are directed to stand and walk 3 meters to a cone on the floor. They are to round the cone in a continuous motion, walk back to the chair, turn again and be seated. The entire test is performed at a comfortable and safe speed for the patient. The data are captured by an Attitude and Heading Reference System (AHRS). Custom software has been developed to appropriately filter the raw data, establish a fixed global coordinate system (i.e. aligned with the body coordinate system), segregate gait segment data from turn data, and delineate and compile data for left and right strides for separate analyses.
Performance test - Five time sit to stand test | 3, 6, 12 months
  Participants begin from a seated position and are directed to come to a full standing position without push off assistance from upper extremities and then return to a seated position without upper extremity assist. The test pattern is repeated 5 times. The data are captured by an Attitude and Heading Reference System (AHRS) that is chest-mounted and positioned at the top of the sternum using a simple harness. Custom software has been developed to appropriately filter the raw data, establish a fixed global coordinate system (i.e. aligned with the body coordinate system), segregate gait segment data from turn data, and delineate and compile data for left and right strides for separate analyses.
Performance test - 10 meter walk test (Gait) | 3, 6, 12 months
  Participants complete a modified 10 meter walk test which involves the subject starting from a standing position, walking 5 meters at a comfortable pace, turning around, and then walking back 5 meters to the original starting point. The test is repeated twice for each subject. The data are captured by an Attitude and Heading Reference System (AHRS) that is chest-mounted and positioned at the top of the sternum using a simple harness. Custom software has been developed to appropriately filter the raw data, establish a fixed global coordinate system (i.e. aligned with the body coordinate system), segregate gait segment data from turn data, and delineate and compile data for left and right strides for separate analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hsu, MD, Principal Investigator — Wake Forest University Health Sciences